CLINICAL TRIAL: NCT03408158
Title: Multi-center Study in the Frequency of HPA Antibodies and the Distribution of Antigen and Antibodies in Chinese Blood Disease Patients
Brief Title: HPA Antibodies and the Distribution of Antigen and Antibodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou First People's Hospital (Other)
Collaborators: LanZhou University (Other); First Affiliated Hospital of Harbin Medical University (Other); Hunan Provincial People's Hospital (Other); The Fourth Affiliated Hospital of China Medical University (Other); The Third Affiliated Hospital of Guangzhou Medical University (Other); First Affiliated Hospital Xi'an Jiaotong University (Other); Nanfang Hospital, Southern Medical University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: K2016-116-01
Record Dates: First submitted 2017-12-04; First posted 2018-01-23 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2019-01

CONDITIONS: Blood Disease; Platelet Refractoriness; Antibody-mediated Rejection
Keywords: HPA; Blood disease
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HPA antigen and antibodies (No Intervention): Investigate the positive rate of HPA antibodies, the distribution and the specificity of HPA antigen and antibodies in Chinese blood disease patients.
- necessity of HPA antibodies screening (No Intervention): Investigate the connection between times of platelet transplantation and HPA antibody titer, which providing statistical data for evaluating the necessity and setting screening time and standards of HPA antibodies screening.
- matched platlet infusion (Experimental): Enable platelet donors'common HPA antigen to be typed and blood disease patients to be same type infusion of main HPA antigen as possible as early.The investigators compare the differences of platelet count between patients with same type infusion of main HPA antigen and not.
  Interventions: Procedure: same type infusion of main HPA antigen

INTERVENTIONS:
Procedure: same type infusion of main HPA antigen — Compare the differences of platelet count between participants with same type infusion of main HPA antigen and not
  Arms: matched platlet infusion

SUMMARY:
By detecting platelet antibodies of participants and then further to identify their genotype and analyzing laboratory examination, the investigators will obtain positive frequency of HPA antibodies, the distribution of HPA antigen and antibodies, effect of matching platelet transfusion, all of which in favor of draw a conclusion that it is very important to carry out HPA antibody detection and matching transfusion in early phase.

DETAILED DESCRIPTION:
1. The investigators will detect platelet antibodies of participants who are according with the inclusive criteria.
2. For participants with platelet antibodies, the investigators should screen out cases owning HPA antibodies and further to identify their genotype.
3. Platelet infusion of same type will be applied to half of participants with HPA antibodies as experimental group, and the another half of participants with hematopathy will be infused ordinary platelets as control. The investigators will estimate the effect of matching transfusion through laboratory examination such as platelet count 1 hour and 24 hours after transfusion and clinical feature comparing to control group.
4. Finally, the investigators will obtain several conclusions includes positive frequency of HPA antibodies, the distribution of HPA antigen and antibodies, effect of matching platelet transfusion by analyzing a bunch of relevant information. So, strong evidence will be provide to decide if it is very important to carry out HPA antibody detection and matching transfusion in early phase.

ELIGIBILITY:
Inclusion Criteria:

1. Blood disease patients with voluntary participation in creating records, no gender limitation, 0-99 years of age, first diagnosed or be hospitalized in our hospital with platelet transfusion more than once.
2. Patients transfers from other hospitals which can be confirm the time (>1) of platelet transfusion.
3. Patient be cured, discharged or dead with the time of platelet transfusion is between 1 to 10 should be included.
4. Patient with HPA antibodies at admission could be considered to be included into same type transfusion group.

   -

Exclusion Criteria:

1. Patients informed but refuse to participate in;
2. Patients with HPA antibodies quitting therapy or breaking off cooperation during research;
3. Patients with many referrals and the time of platelet transfusion can not be confirmed;
4. Patient without platelet transfusion;
5. Patient with termination of treatment whatever active or passive. -

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6170 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
The percentages (%) of hematopoietic patients with anti-HPA antibodies among all investigated hematopoietic patients who need long-term infusion of platelets. | From one participant first enrolled in this study to the moment of HPA antibodies could be detected or death, up to 6 months. The investigators will calculate the percentages after all participants are done with trace.
  The investigators will recruit about 25000 participants in total (anticipated) of different hospitals spread over the whole country and divide them into two categories, patients with and patients without platelet antibodies, by detecting antibodies through solid-phase agglutination (qualitative analysis). The investigators screen out the positive ones and then distinguish participants with antibodies against human platelet antigens (HPA) from those with antibodies against human leukocyte antigens (HLA) by using LIFECODES PAKPLUS (qualitative analysis). At the same time, subtype of anti-HPA antibodies (such as anti-HPA-1a antibodies) are detected. The analyzation of large sample data will present investigators the most important findings, the percentages (%, the primary outcome measure) of hematopoietic patients with anti-HPA antibodies (include the total and the various subtypes) among all investigated hematopoietic patients who need long-term infusion of platelets.

CONTACTS AND LOCATIONS:
Overall Officials: Yaming Wei, Doctor, Study Chair — Director of Blood Transfusion Department
Locations (1):
- Guangzhou First People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
We plan to share IPD with other researchers 5 years after the termination of the whole study.

REFERENCES:
- [Background] Berry J, Allen D, Porcelijn L, de Haas M, Kekomaki R, Kaplan C, Ouwehand WH, Metcalfe P. Collaborative studies to establish the first World Health Organization International Standard for detection of human antibody against human platelet antigen-3a. Vox Sang. 2007 Nov;93(4):309-15. doi: 10.1111/j.1423-0410.2007.00899.x. PMID 18070275
- [Background] Kerkhoffs JL, Eikenboom JC, van de Watering LM, van Wordragen-Vlaswinkel RJ, Wijermans PW, Brand A. The clinical impact of platelet refractoriness: correlation with bleeding and survival. Transfusion. 2008 Sep;48(9):1959-65. doi: 10.1111/j.1537-2995.2008.01799.x. Epub 2008 Jun 28. PMID 18564396
- [Background] Meehan KR, Matias CO, Rathore SS, Sandler SG, Kallich J, LaBrecque J, Erder H, Schulman KA. Platelet transfusions: utilization and associated costs in a tertiary care hospital. Am J Hematol. 2000 Aug;64(4):251-6. doi: 10.1002/1096-8652(200008)64:43.0.co;2-n. PMID 10911376
- [Background] Mishima Y, Tsuno NH, Matsuhashi M, Yoshizato T, Sato T, Ikeda T, Watanabe-Okochi N, Nagura Y, Sone S, Kurokawa M, Okazaki H. Effects of universal vs bedside leukoreductions on the alloimmunization to platelets and the platelet transfusion refractoriness. Transfus Apher Sci. 2015 Feb;52(1):112-21. doi: 10.1016/j.transci.2014.11.001. Epub 2014 Nov 11. PMID 25467707
- [Background] Ramirez P, Brunstein CG, Miller B, Defor T, Weisdorf D. Delayed platelet recovery after allogeneic transplantation: a predictor of increased treatment-related mortality and poorer survival. Bone Marrow Transplant. 2011 Jul;46(7):981-6. doi: 10.1038/bmt.2010.218. Epub 2010 Oct 4. PMID 20921943
- [Background] Macher S, Schallmoser K, Staber PB, Neumeister P, Posch U, Lanzer G, Panzer S. Severe thrombocytopenia due to host-derived anti-HPA-1a after non-myeloablative allogeneic haematopoietic stem cell transplantation for multiple myeloma: a case report. Vox Sang. 2005 Nov;89(4):257-60. doi: 10.1111/j.1423-0410.2005.00692.x. PMID 16262760
- [Background] Lucas G, Culliford S, Green F, Sidra G, Calvert A, Green A, Harrison P, Harvey J, Allen D, Smillie D, Masurekar A, Marks D, Russell N, Massey E. Recipient-derived HPA-1a antibodies: a cause of prolonged thrombocytopenia after unrelated donor stem cell transplantation. Transfusion. 2010 Feb;50(2):334-9. doi: 10.1111/j.1537-2995.2009.02448.x. Epub 2009 Oct 23. PMID 19874563